CLINICAL TRIAL: NCT04704414
Title: Exophthalmometry With 3D Face Scanners
Acronym: EX3D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Konrad Peter Weber, Principal Investigator, University of Zurich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BASEC-Nr. 2019-00233; CIV-19-08-029404 (Other: EUDAMED); 10000520 (Other: Swissmedic)
Record Dates: First submitted 2021-01-06; First posted 2021-01-11 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Exophthalmos; Graves Ophthalmopathy; Orbital Tumor; Orbital Fractures
Keywords: Hertel exophthalmometer; exophthalmos; face scanner; smartphone
MeSH Terms: conditions — Exophthalmos; Graves Ophthalmopathy; Orbital Neoplasms; Orbital Fractures

STUDY DESIGN:
Intervention Model Description: * Accuracy and precision of smartphone in comparison with 3D face scanner and Hertel exophthalmometer
  * Test-retest reliability
  * Inter-operator reliability
  * Before and after exophthalmos-changing intervention
Masking Description: Blinding of the operators of Hertel exophthalmometer for previous measurement results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Validation of smartphone face scanner (Experimental): Validation of smartphone face scanner in comparison to Hertel Exophthalmometer and high-definition face scanner.
  Interventions: Device: Exophthalmos measurement

INTERVENTIONS:
Device: Exophthalmos measurement — Exophthalmos measurement with iPhone 11 vs Artec Space Spider 3D Scanner vs Hertel Exophthalmometer.

SUMMARY:
This study investigates diagnostic methods to measure eyeball protrusion with a smartphone face scanner compared to the traditional Hertel exophthalmometer. The study aims to validate a new reliable, fast and convenient smartphone app to measure the protrusion of the eyeball in different diseases such as Graves' disease, orbital tumors, orbital fractures or orbital inflammation, as well as other rare diseases.

DETAILED DESCRIPTION:
BACKGROUND: Accurate and reproducible measures of abnormal eyeball protrusion are important for diagnosing different causes of exophthalmos, as well as following patients with Grave's orbitopathy and retroorbital tumors. The current clinical gold standards for measuring abnormal eyeball protrusion is the Hertel exophthalmometer, which is prone to reading errors and inconvenient to use.

OBJECTIVE: The purpose of the EX3D-project is to replace the historic Hertel Exophthalmometer with a state-of-the-art mobile smartphone app that every ophthalmologist can carry in his pocket.

METHODS: The investigators developed an accurate and easy to use method for measuring abnormal eyeball protrusion using the TrueDepth camera of the iPhone 11 in comparison with a high-resolution 3D scanner as a reference to compare with the Hertel Exophthalmometer.

OUTCOMES:

1. Accuracy and precision of 3D face-scanner and iPhone in comparison to Hertel Exophthalmometer.
2. Test re-test reliability in comparison to Hertel Exophthalmometer.
3. Inter-operator reliability against Hertel Exophthalmometer.
4. Patients before and after exophthalmos changing treatment.
5. Applicability in daily clinical practice.

BROADER IMPACT: The invention makes exophthalmometry quick, easy and objective. A mobile smartphone application would replace measurements with the traditional Hertel Exophthalmometer, which are cumbersome, prone to reading errors and have a poor inter-rater reliability as well as test-retest reliability.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Able to cooperate with the study investigations (hearing, comprehension)
* Exophthalmos (Grave's disease, orbital tumors, orbital inflammation, orbital fractures, rare causes (congenital, e.g. microphthalmos)
* health controls

Exclusion Criteria:

* Unable to sign informed consent
* Unable to cooperate with the examinations (hearing loss, neurological deficits)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-08-14 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the smartphone face scanner | On average 2 weeks
  Accuracy of iPhone exophthalmos measurements (measured in mm for each eye) compared to measure with 3D face scanner and Hertel Exophthalmometer
Test-retest-reliability of the smartphone face scanner | On average 2 weeks
  Repeated measures (measured in mm for each eye) of the same subjects with iPhone 11, Hertel Exophthalmometer and 3D face scanner
Inter-operator reliability of the smartphone face scanner | On average 2 weeks
  Measurement (measured in mm for each eye) of the same patients by 3 different operators
Smartphone face scanner measures before and after treatment with the smartphone face scanner | On average 3 months
  Measurements (measured in mm for each eye) with the smartphone face scanner before and after exophthalmos-changing treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmology Department, University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided